CLINICAL TRIAL: NCT02001740
Title: Treatment of Adhesive Capsulitis: A Randomized Placebo-Controlled Trial Comparing Arthrographic Joint Distention With Steroid and Local Anesthetic Versus Arthrographic Joint Distention With Local Anesthetic Alone
Brief Title: An RCT in Treatment of Adhesive Capsulitis Arthrographic Joint Distention With Local Anesthetic Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Ryan Bicknell, Assistant Professor, Queen's University., Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SURG-246-12
Record Dates: First submitted 2013-08-20; First posted 2013-12-05 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Adhesive Capsulitis
Keywords: shoulder
MeSH Terms: conditions — Bursitis | interventions — Steroids; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- lidocaine (Placebo Comparator): frequency = once
  Interventions: Other: Lidocaine
- Triamcinalone (steroid) and lidocaine (Experimental): frequency = once
  Interventions: Drug: Triamcinalone (steroid) and lidocaine

INTERVENTIONS:
Drug: Triamcinalone (steroid) and lidocaine — receive once
  Arms: Triamcinalone (steroid) and lidocaine
Other: Lidocaine — receive once
  Arms: lidocaine

SUMMARY:
Frozen shoulder or adhesive capsulitis is a common cause of shoulder pain, estimated to affect 25% of the general population. Many forms of treatment have been advocated for frozen shoulder including physiotherapy, injection with steroid, distension arthrogram with steroid, manipulation under anesthetic and arthroscopic releases. There is no general agreement in favour of one form of treatment, and the response to a particular treatment varies in different series. A few randomized controlled trials appear in the literature. Most of these showed improvements with steroid use, but the results were not always statistically significant. One randomized control trial reported superior results in favor of arthrographic joint distension with steroid compared to a saline placebo. To our knowledge there have been no other similar randomized trials to support these results. The objective of this study is to determine if arthrographic distension of the shoulder joint with steriods is an effective treatment modality for adhesive capsulitis as compared to injection with local anesthetic and contrast alone. The study design is a placebo-controlled, double blind clinical trial where participants will undergo distension arthrogram of the shoulder and be randomized to receive either Triamcinalone (steroid), lidocaine and contrast or injection with lidocaine and contrast alone.

ELIGIBILITY:
Inclusion Criteria:

* Age range 19-70
* Female and male
* Ability to understand and give consent
* Diagnosis of adhesive capsulitis (frozen shoulder) pain and stiffness for at least 3 months.

Exclusion Criteria:

* • Frozen shoulder secondary to trauma

  * Previous surgery on the affected shoulder
  * Age less than 19 or greater than 70
  * Systemic inflammatory joint disease such as Rheumatoid Arthritis
  * Radiographic evidence of osteoarthritis of the shoulder
  * Allergy to contrast material
  * Pregnant or breastfeeding women

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
functional outcomes as determined by the SPADI | change in baseline at 1 year.

SECONDARY OUTCOMES:
passive range of motion | baseline, 3 and 6 and 12 week post injection.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bicknell, MD, Principal Investigator — Queen's University and Kingston General Hospital
Locations (1):
- Kingston General and Hotel Dieu Hospitals, Kingston, Ontario, Canada